CLINICAL TRIAL: NCT00143598
Title: The SOX Trial: Compression Stockings to Prevent the Post-Thrombotic Syndrome After Symptomatic Proximal Deep Venous Thrombosis
Brief Title: The SOX Trial: Compression Stockings to Prevent the Post-Thrombotic Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Sigvaris Corporation (Industry)
Responsible Party: Principal Investigator, Dr. Susan Kahn, SOX Trial Principal Investigator, Sir Mortimer B. Davis - Jewish General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MCT-63142; ISRCTN71334751 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Results first posted 2014-08-18 (Estimated); Last update posted 2014-08-18 (Estimated); Status verified 2014-08

CONDITIONS: Deep Venous Thrombosis
Keywords: Postphlebitic Syndrome; Post-Thrombotic Syndrome; Elastic Stockings; Stockings, Compression; Randomized Controlled Trials; Quality of Life
MeSH Terms: conditions — Venous Thrombosis; Postphlebitic Syndrome; Postthrombotic Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active ECS (Active Comparator): Active Elastic Compression Stockings (ECS) 30-40 mm Hg compression at the ankle.
  Interventions: Device: Knee-length, graduated elastic compression stocking
- Placebo ECS (Placebo Comparator): Placebo stockings with identical appearance to Active ECS and with < 5 mm Hg compression at the ankle.
  Interventions: Device: Knee-length, placebo stocking

INTERVENTIONS:
Device: Knee-length, graduated elastic compression stocking — Worn daily for 2 years, 30-40 mm Hg
  Arms: Active ECS
Device: Knee-length, placebo stocking — Worn daily for two years
  Arms: Placebo ECS

SUMMARY:
The purpose of this study is to determine whether elastic compression stockings used for 2 years are effective in preventing the post-thrombotic syndrome in patients with symptomatic proximal deep venous thrombosis.

DETAILED DESCRIPTION:
The post-thrombotic syndrome (PTS) is a frequent, burdensome and costly condition that occurs in about one third of patients after an episode of deep vein thrombosis (DVT). Affected patients have chronic leg pain and swelling, and sometimes develop skin ulcers. At present, there is little to offer for the treatment of this condition. Prevention of PTS is the key to reducing its burden on patients and society. Elastic compression stockings (ECS) could be helpful in preventing PTS, however data on their effectiveness are scarce and conflicting.

Comparison(s): Knee-length, 30-40 mm Hg (Class II), graduated ECS worn on the DVT-affected leg daily for 2 years compared to knee-length, inactive (i.e. no compression) stocking, identical in appearance to active ECS, worn on the DVT-affected leg daily for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with a first, symptomatic, objectively confirmed proximal DVT diagnosed within the last 14 days (with or without concurrent distal DVT or pulmonary embolism)
* Who have no contraindications to standard treatment with heparin and/or warfarin, and
* Who provide informed consent to participate

Exclusion Criteria:

* Contraindication to compression stockings
* Limited lifespan (estimated < 6 months)
* Geographic inaccessibility preventing return for follow-up visits
* Inability to apply stockings daily and unavailability of a caregiver to apply stockings daily
* Treatment of acute DVT with thrombolytic agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 806 (Actual)
Dates: Start 2004-06; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan R. Kahn, M.D., M.Sc., Principal Investigator — Sir Mortimer B. Davis - Jewish General Hospital
Locations (25):
- United States (3):
  - Henry Ford Health Systerm, Detroit, Michigan
  - Duke University Medical Center, Durham, North Carolina
  - Oklahoma University Health Sciences Center, Oklahoma City, Oklahoma
- Canada (22):
  - Victoria Heart Institute Foundation, Victoria, British Columbia
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - QE II Health Sciences Centre, Halifax, Nova Scotia
  - Hamilton Health Sciences - General Hospital, Hamilton, Ontario
  - Hamilton Health Sciences - Chedoke Division, Hamilton, Ontario
  - Hamilton Health Sciences - McMaster University Medical Centre, Hamilton, Ontario
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Hamilton Health Sciences - Henderson General Hospital, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - The Ottawa Hospital, Civic Campus, Ottawa, Ontario
  - Sunnybrook & Women's College Health Sciences Centre, Toronto, Ontario
  - University Health Network - Toronto General Hospital, Toronto, Ontario
  - Centre Hospitalier Pierre-Boucher, Longueuil, Quebec
  - Hôpital Maisonneuve-Rosemont, Montreal, Quebec
  - Centre Hospitalier de l'Université de Montréal - Hôpital Notre-Dame, Montreal, Quebec
  - Centre Hospitalier de l'Université de Montréal - Hôpital Hôtel-Dieu, Montreal, Quebec
  - Royal Victoria Hospital - McGill University Health Centre, Montreal, Quebec
  - Sir Mortimer B. Davis - Jewish General Hospital, Montreal, Quebec
  - St. Mary's Hospital Center, Montreal, Quebec
  - Montreal General Hospital - McGill University Health Centre, Montreal, Quebec
  - Hôpital du Sacré-Coeur de Montréal, Montreal, Quebec
  - Centre hospitalier affilié universitaire de Québec, Hôpital de l'Enfant-Jésus, Québec, Quebec

REFERENCES:
- [Background] Kahn SR, Shbaklo H, Shapiro S, Wells PS, Kovacs MJ, Rodger MA, Anderson DR, Ginsberg JS, Johri M, Tagalakis V; SOX Trial Investigators. Effectiveness of compression stockings to prevent the post-thrombotic syndrome (the SOX Trial and Bio-SOX biomarker substudy): a randomized controlled trial. BMC Cardiovasc Disord. 2007 Jul 24;7:21. doi: 10.1186/1471-2261-7-21. PMID 17711595
- [Result] Kahn SR, Shapiro S, Wells PS, Rodger MA, Kovacs MJ, Anderson DR, Tagalakis V, Houweling AH, Ducruet T, Holcroft C, Johri M, Solymoss S, Miron MJ, Yeo E, Smith R, Schulman S, Kassis J, Kearon C, Chagnon I, Wong T, Demers C, Hanmiah R, Kaatz S, Selby R, Rathbun S, Desmarais S, Opatrny L, Ortel TL, Ginsberg JS; SOX trial investigators. Compression stockings to prevent post-thrombotic syndrome: a randomised placebo-controlled trial. Lancet. 2014 Mar 8;383(9920):880-8. doi: 10.1016/S0140-6736(13)61902-9. Epub 2013 Dec 6. PMID 24315521
- [Derived] Kahn SR, Shapiro S, Ducruet T, Wells PS, Rodger MA, Kovacs MJ, Anderson D, Tagalakis V, Morrison DR, Solymoss S, Miron MJ, Yeo E, Smith R, Schulman S, Kassis J, Kearon C, Chagnon I, Wong T, Demers C, Hanmiah R, Kaatz S, Selby R, Rathbun S, Desmarais S, Opatrny L, Ortel TL, Galanaud JP, Ginsberg JS. Graduated compression stockings to treat acute leg pain associated with proximal DVT. A randomised controlled trial. Thromb Haemost. 2014 Dec;112(6):1137-41. doi: 10.1160/TH14-05-0430. Epub 2014 Aug 28. PMID 25183442
- See also: Biomarker Sub Study of the Compression Stockings to Prevent the Post-Thrombotic Syndrome (SOX) Trial (Bio-SOX) — http://clinicaltrials.gov/ct2/show/NCT01615705

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between June, 2004, and February, 2010, we enrolled patients in 24 centres in Canada and the USA.
Pre-assignment Details: Patients were excluded if they had a contraindication to the use of compression stockings, an expected life span of <6 months, geographical inaccessibility, were unable to apply stockings, or received thrombolytic therapy for the initial treatment of acute deep vein thrombosis (DVT).
Groups:
- Active ECS: Active Elastic Compression Stockings. 30-40 mm Hg
- Placebo ECS: Placebo stockings with identical appearance but less than 5 mm Hg compression at the ankle.
Period: Overall Study
Arm/Group | Active ECS | Placebo ECS
Started | 410 | 396
Completed | 318 | 302
Not Completed | 92 | 94
Not completed — Lost to Follow-up | 23 | 21
Not completed — Withdrawal by Subject | 33 | 37
Not completed — Death | 36 | 36

BASELINE CHARACTERISTICS:
Population: 806 patients were randomly assigned to an intervention. Three patients were identified as ineligible soon after randomization and were excluded from further analysis (ie, modified intention-to-treat). In the active ECS group, one patient had no DVT and in the placebo ECS group one patient had a previous DVT and another patient was moribund.
Groups:
- Total: Total of all reporting groups
Arm/Group | Active ECS | Placebo ECS | Total
Number analyzed (Participants) | 409 | 394 | 803
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (15.3) | 54.8 (15.8) | 55.1 (15.5)
Age, Customized [Number; unit: participants]
  <40 years | 67 | 67 | 134
  40-65 years | 222 | 217 | 439
  >65 years | 120 | 110 | 230
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 154 | 166 | 320
  Male | 255 | 228 | 483
Race/Ethnicity, Customized [Number; unit: participants]
  White ethnic origin | 371 | 354 | 725
Outpatients [Number; unit: participants] | 355 | 344 | 699
Body-mass index, kg/m2 [Mean (Standard Deviation); unit: kg/m^2] | 29.0 (6.1) | 28.9 (6.1) | 28.95 (6.1)
Time from DVT diagnosis to randomization [Mean (Standard Deviation); unit: days] | 4.8 (4.1) | 4.6 (3.8) | 4.7 (3.9)
Side of DVT [Number; unit: participants]
  Left | 180 | 173 | 353
  Right | 222 | 216 | 438
  Bilateral | 7 | 5 | 12
Most proximal extent of DVT [Number; unit: participants]
  Iliac vein | 44 | 49 | 93
  Common femoral vein | 109 | 107 | 216
  Femoral Vein | 128 | 123 | 251
  Popliteal vein | 128 | 115 | 243
Villalta score at baseline [Mean (Standard Deviation); unit: Score on a scale] — The Villalta Scale for assessment of the post-thrombotic syndrome
  The Villalta scale has a range of 0-33. A Villalta scale score >4 indicates post-thrombotic syndrome (severity of post-thrombotic syndrome is categorized as 5-9 points, mild; 10-14 points, moderate; >14 points or presence of an ulcer, severe).
  Higher values signify worse outcome.
  Points on each item in the scale are simply summed to a total score.
  Score on a scale | 8.2 (4.4) | 8.7 (4.8) | 8.4 (4.6)
Concurrent pulmonary embolism [Number; unit: participants] | 57 | 57 | 114
Venous thrombosis risk factors [Number; unit: participants]
  Surgery, past 3 months | 77 | 64 | 141
  Trauma, past 3 months | 42 | 51 | 93
  Immobilised in past month | 67 | 61 | 128
  Active cancer | 52 | 46 | 98
  Pregnant, post partum, OCT, or HRT | 37 | 55 | 92
  Family history of venous thromboembolism | 85 | 82 | 167
Type of DVT Treatment [Number; unit: participants]
  Low molecular weight heparin | 388 | 384 | 772
  Unfractionated heparin | 31 | 21 | 52
  Warfarin | 330 | 317 | 647
  Investigational anitcoagulant | 15 | 11 | 26
Duration of DVT Treatment [Median (Inter-Quartile Range); unit: days]
  Duration of heparin | 8 [6 to 11] | 8 [6 to 10] | 8 [6 to 11]
  Duration of Oral Anti-Coagulation (OAC) | 186 [113 to 253] | 182 [104 to 220] | 185 [109.5 to 231]

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Post-thrombotic Syndrome (PTS)
Time Frame: During 2-year follow up
Population: Intention to treat.
Measure: Number; unit: participants
Arm/Group | Active ECS | Placebo ECS
Number analyzed (Participants) | 409 | 394
participants | 44 | 37
Statistical Analysis 1: Comparison: Active ECS vs Placebo ECS; Test type: Superiority or Other; p = .58, Regression, Cox; Adjusted for centre; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [.73 to 1.76]

2. Secondary Outcome: Severity of PTS, Including Incidence of Venous Ulcer
Description: Highest Villalta at or after 6 month visit
  The Villalta Scale for assessment of the post-thrombotic syndrome The Villalta scale has a range of 0-33. A Villalta scale score >4 indicates post-thrombotic syndrome (severity of post-thrombotic syndrome is categorized as 5-9 points, mild; 10-14 points, moderate; >14 points or presence of an ulcer, severe).
  Higher values signify worse outcome. Points on each item in the scale are simply summed to a total score.
Time Frame: 6-24 months.
Population: Highest Villalta score at or after 6 month visit (missing for 48 patients in each group).
Measure: Number; unit: participants
Arm/Group | Active ECS | Placebo ECS
Number analyzed (Participants) | 361 | 346
participants
  None (score <5) | 185 | 178
  Mild (5-9) | 119 | 111
  Moderate (10-14) | 30 | 37
  Severe (>14 or ulcer) | 27 | 20

3. Secondary Outcome: Incidence of Objectively Confirmed Recurrent Venous Thromboembolism (VTE), Death From VTE and Major Bleeding
Time Frame: During 2-year follow up
Measure: Number; unit: participants
Arm/Group | Active ECS | Placebo ECS
Number analyzed (Participants) | 409 | 394
participants
  Recurrent venous thromboembolism | 33 | 38
  Death from VTE | 0 | 0
  Major bleeding | 11 | 14

4. Secondary Outcome: Quality of Life
Description: The SF-36 is a well-validated generic quality-of-life (QOL) instrument. It includes questions on both physical and mental health. Higher scores indicate a better QOL. The VEINES-QOL is a venous-disease specific QOL measure that consists of 25 items that quantify venous disease effect on QOL, and an embedded symptom sub-questionnaire (VEINES-Sym) with 10 items that measures venous symptoms. Higher scores are associated with better QOL.
  The VEINES-QOL/Sym and SF-36 use the standard method for scoring questionnaires with items with different response scales that is now routinely used. Raw scores are first transformed to z score equivalents (mean, 0; standard deviation, 1), which then are transformed to T scores (mean, 50; standard deviation, 10) to give an easily understood range of scores. A person-specific estimate is imputed for any missing item in cases where the patient answered at least 50% of the items in the scale.
Time Frame: 24 months
Population: Patients who completed the SF-36 and VEINES-QOL at 24 months follow-up.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Active ECS | Placebo ECS
Number analyzed (Participants) | 268 | 261
Scores on a scale
  SF-36 PCS | 46.7 (10.7) | 47.5 (10.2)
  SF-36 MCS | 52.7 (9.3) | 52.5 (8.8)
  VEINES-QOL | 56.6 (5.3) | 57.4 (5.3)

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Active ECS | Placebo ECS
Serious Adverse Events (participants affected / at risk) | 0/409 | 0/394
Other Adverse Events (participants affected / at risk) | 8/409 | 7/394
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active ECS (N=409) | Placebo ECS (N=394)
Rash/Itching (Skin and subcutaneous tissue disorders) | 8 (8) | 7 (7)

LIMITATIONS AND CAVEATS:
While 14% withdrew or were lost to follow-up (F/U), the total rate of withdrawal, loss to F/U and death was less than what was projected. Adherence to study stockings tended to diminish over F/U; this occurred to a similar degree in both groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No